CLINICAL TRIAL: NCT05183867
Title: Comparing the Healthy Minds Program With an Active Control and Waitlist Control in Depression
Brief Title: Behavior, Biology and Well-Being Study
Acronym: BeWell
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Hope for Depression Research Foundation (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-0991; Protocol Version 6/29/2023 (Other: UW Madison); A487400 (Other: UW Madison); 1U24AT011289-01 (NIH)
Record Dates: First submitted 2021-12-21; First posted 2022-01-11 (Actual); Results first posted 2025-08-01 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Depression; Psychological Distress
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: The groups will be randomized to one of three groups in a 2:2:1 ratio.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy Minds Program (HMP) app (Experimental): Participants will receive access to the 4-week HMP Foundations module. The HMP app is a meditation-based smartphone app designed to promote and protect psychological well-being through sustainable skills training. The program is grounded in constituents of psychological well-being identified in empirical literature. HMP provides core content, with instruction administered through a curriculum of guided practices. HMP is based on research on eudaimonic well-being (e.g., environmental mastery, purpose) and brain-based skills that underlie these qualities (e.g., regulation of attention, mental flexibility). The full HMP has guided audio practices that address 4 constituents of well-being: awareness, connection, insight, and purpose. At post-treatment, participants will be given access to additional HMP content to support their continued practice.
  Interventions: Device: Healthy Minds Program
- Psychoeducation app (Active Comparator): Participants will receive access to the 4-week HMP Foundations module with guided meditation practices removed. The active control will include only the didactic content included in HMP without the guided meditation practices.
  Interventions: Device: Healthy Minds Program
- Usual Care (No Intervention): Participants will receive access to HMP at the end of the study and will be encouraged to continue with their usual care.

INTERVENTIONS:
Device: Healthy Minds Program — HMP is a 4-week mobile health (mHealth) meditation training program.
  Other Names: HMP
  Arms: Healthy Minds Program (HMP) app; Psychoeducation app

SUMMARY:
The central aim of this study is to test the efficacy of the Healthy Minds Program (HMP) app, an intervention designed to promote well-being. The investigators plan to conduct a randomized controlled trial (RCT) involving 1100 participants comparing 4-weeks of the HMP app with an active control (Psychoeducation [HMP without meditation practice]), and a waitlist control in a sample of United States adults with elevated depression symptoms.

DETAILED DESCRIPTION:
Depression is highly prevalent and associated with extreme personal and societal costs. Meditation training reduces depression symptoms and psychological distress, but access to in-person programs is limited due to associated cost and lack of available services. Research on neurocognitive and biological mechanisms of meditation training in alleviating depression is at a preliminary stage, and an obstacle limiting research progress is over-reliance on retrospective self-report measures, which are vulnerable to a host of biases. This project will use gold-standard behavioral measures and explore novel measures of relevant neurocognitive and behavioral processes, namely pattern separation, self-referential thought, and video-based assessment of emotional well-being. Furthermore, the project will investigate effects on the gut microbiome (with fecal samples) and inflammation (with dried blood spots), which reflect biological systems hypothesized to be mechanistically related to benefits of meditation and well-being training.

ELIGIBILITY:
Inclusion Criteria:

* Elevated PHQ-8 or PHQ-9 ≥ 5 at screening
* Proficient in English
* Able to provide informed consent
* Have access to a smartphone that can download apps from Google Play or the Apple App Store
* For payment purposes, must be a US citizen or a permanent US resident

Exclusion Criteria:

* Regular daily meditation practice for past 6 months or regular weekly meditation practice for past 12 months
* Attended a meditation retreat or a yoga/body practice retreat with a significant meditation component

  - Previous use of Healthy Minds Program app
* Current suicidal intent and/or high self-injury risk (determined from the interview)
* Self-reported history of psychosis
* Self-reported history of mania
* Current psychopathology that interferes with study participation as assessed by interview
* Living or traveling outside the US during the whole study participation period (trips outside US after the interview phase is not an exclusion)
* Alcohol Use Disorders Identification Test (AUDIT) score ≥ 13 for women and AUDIT score ≥ 15 for men
* Drug Use Disorders Identification Test (DUDIT) score ≥ 8 for women and men

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1157 (Actual)
Dates: Start 2022-03-24 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simon Goldberg, PhD, Principal Investigator — UW-Madison, Center for Healthy Minds
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care
Started | 462 | 463 | 232
Completed | 459 | 461 | 232
Not Completed | 3 | 2 | 0
Not completed — Withdrawal by Subject | 3 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care | Total
Number analyzed (Participants) | 462 | 463 | 232 | 1157
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.34 (11.84) | 39.02 (12.18) | 38.72 (12.64) | 38.69 (12.13)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Man | 93 | 103 | 49 | 245
  Woman | 355 | 342 | 173 | 870
  Other | 3 | 7 | 2 | 12
  Unknown or Not Reported | 11 | 11 | 8 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 48 | 40 | 24 | 112
  Not Hispanic or Latino | 400 | 406 | 198 | 1004
  Unknown or Not Reported | 14 | 17 | 10 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 5 | 1 | 8
  Asian | 26 | 24 | 12 | 62
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1 | 2
  Black or African American | 36 | 46 | 21 | 103
  White | 341 | 357 | 176 | 874
  More than one race | 45 | 25 | 12 | 82
  Unknown or Not Reported | 12 | 5 | 9 | 26
Region of Enrollment [Number; unit: participants]
  United States | 462 | 463 | 232 | 1157

OUTCOME MEASURES:

1. Primary Outcome: Depression Symptoms Measured by Patient Health Questionnaire - 8 (PHQ-8) Score
Description: The PHQ-8 is an 8-item questionnaire where participants report how often in the past 2 weeks they were bothered by specific problems. It is scored on a 4-point Likert scale where 0 = not at all to 3 = nearly every day. The total possible range of scores is 0-24 where higher scores indicate more depressive symptoms.
Time Frame: Baseline, week 1, week 2, week 3, week 4 (of intervention period), and 3 month follow-up
Population: Some participants did not provide data at all time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Healthy Minds Program (HMP) App: Participants will receive full access to the 4-week HMP Foundations module. The full HMP has guided audio practices that address 4 constituents of well-being: awareness, connection, insight, and purpose. At post-treatment, participants will be given access to additional HMP content to support their continued practice.
  Healthy Minds Program: HMP is a 4-week mobile health (mHealth) meditation training program.
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care
Number analyzed (Participants) | 462 | 463 | 232
score on a scale
  baseline | 10.06 (4.85) | 9.85 (4.68) | 9.79 (4.75)
  Week 1: number analyzed (Participants) | 403 | 407 | 216
  Week 1 | 9.17 (4.72) | 8.8 (4.71) | 9.45 (5.11)
  Week 2: number analyzed (Participants) | 376 | 377 | 204
  Week 2 | 8.37 (4.75) | 8.28 (4.6) | 9.03 (5.22)
  Week 3: number analyzed (Participants) | 372 | 366 | 204
  Week 3 | 7.88 (4.9) | 8.01 (4.84) | 9.21 (4.93)
  Week 4: number analyzed (Participants) | 395 | 389 | 218
  Week 4 | 7.21 (4.8) | 7.39 (4.8) | 8.86 (5.11)
  3-month follow-up: number analyzed (Participants) | 374 | 369 | 204
  3-month follow-up | 6.67 (4.6) | 6.93 (4.92) | 8.46 (5.09)

2. Secondary Outcome: Anxiety Symptoms Measured by Generalized Anxiety Disorder - 7 (GAD-7) Score
Description: The GAD-7 is a 7-item questionnaire where participants report how often in the past 2 weeks they were bothered by specific problems. It is scored on a 4-point Likert scale where 0 = not at all to 3 = nearly every day. The total possible range of scores is 0-21 where higher scores indicate more anxious symptoms.
Time Frame: Baseline, week 1, week 2, week 3, week 4 (of intervention period), and 3 month follow-up
Population: Some participants did not provide data at all time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care
Number analyzed (Participants) | 462 | 463 | 232
score on a scale
  baseline | 8.94 (4.95) | 8.67 (4.97) | 8.37 (4.97)
  Week 1: number analyzed (Participants) | 403 | 407 | 216
  Week 1 | 8.58 (4.88) | 8.13 (4.97) | 8.04 (5.27)
  Week 2: number analyzed (Participants) | 376 | 377 | 204
  Week 2 | 7.66 (4.66) | 7.46 (4.88) | 7.68 (5.04)
  Week 3: number analyzed (Participants) | 372 | 366 | 204
  Week 3 | 7.21 (4.6) | 7.15 (4.71) | 7.59 (5.16)
  Week 4: number analyzed (Participants) | 395 | 389 | 218
  Week 4 | 6.39 (4.55) | 6.46 (4.6) | 7.28 (5.19)
  3-month follow-up: number analyzed (Participants) | 373 | 369 | 204
  3-month follow-up | 6.1 (4.63) | 6.22 (4.75) | 7.08 (5.09)

3. Secondary Outcome: Sleep Disturbance Measured by Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance Score
Description: The PROMIS Sleep Disturbance scale is a computer-adaptive measure where participants report how often in the past 7 days they had various sleep-related experiences (e.g., "my sleep was restful"). It is scored on a 5-point Likert scale where 1 = not at all to 5 = very much. It provides total scores as T-scores (mean = 50, standard deviation (SD) = 10) where higher scores indicate more sleep disturbance.
Time Frame: Baseline, week 1, week 2, week 3, week 4 (of intervention period), and 3 month follow-up
Population: Some participants did not provide data at all time points.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care
Number analyzed (Participants) | 462 | 463 | 232
T-score
  baseline | 57.73 (8.03) | 56.94 (8.16) | 56.9 (8.41)
  Week 1: number analyzed (Participants) | 402 | 407 | 215
  Week 1 | 56.26 (8.35) | 55.91 (8.31) | 57.12 (8.67)
  Week 2: number analyzed (Participants) | 376 | 377 | 204
  Week 2 | 55.78 (8.93) | 55.48 (8.04) | 55.65 (9.19)
  Week 3: number analyzed (Participants) | 371 | 366 | 204
  Week 3 | 55.14 (9.24) | 54.8 (8.96) | 56.53 (8.95)
  Week 4: number analyzed (Participants) | 395 | 389 | 217
  Week 4 | 54.23 (9.06) | 54.17 (8.76) | 55.81 (9.23)
  3-month follow-up: number analyzed (Participants) | 368 | 368 | 201
  3-month follow-up | 53.61 (9.1) | 53.51 (9.29) | 55.76 (9.31)

4. Secondary Outcome: Flourishing Measured by the Flourishing Index Score
Description: The Flourishing Index is a 10-item questionnaire where participants report their general level of flourishing (e.g., well-being, health, etc.). It is scored on a 0 to 10-point scale, with anchors varying across items. The total score ranges from 0 to 100 with higher scores indicating higher flourishing.
Time Frame: Baseline, week 1, week 2, week 3, week 4 (of intervention period), and 3 month follow-up
Population: Some participants did not provide data at all time-points
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care
Number analyzed (Participants) | 462 | 463 | 232
score on a scale
  baseline | 56.26 (15.33) | 56.55 (16.05) | 56.63 (15.22)
  Week 1: number analyzed (Participants) | 404 | 408 | 215
  Week 1 | 57.19 (15.69) | 57.52 (15.83) | 57.22 (14.9)
  Week 2: number analyzed (Participants) | 377 | 377 | 204
  Week 2 | 60.11 (15.58) | 59.92 (15.85) | 58.18 (16.38)
  Week 3: number analyzed (Participants) | 372 | 365 | 204
  Week 3 | 62.45 (15.95) | 60.87 (15.77) | 58.30 (15.80)
  Week 4: number analyzed (Participants) | 395 | 389 | 218
  Week 4 | 64.53 (16.54) | 63.52 (16.42) | 59.29 (16.43)
  3-month follow-up: number analyzed (Participants) | 374 | 369 | 203
  3-month follow-up | 66.00 (16.58) | 64.62 (16.76) | 60.99 (15.43)

5. Secondary Outcome: Awareness Measured by Five Facet Mindfulness Questionnaire Acting With Awareness Subscale Score
Description: The Five Facet Mindfulness Questionnaire Acting with Awareness Subscale is a 8-item subscale where participants report on their general ability to focus. It is scored on a 5-point Likert scale where 1 = never or very rarely true to 5 = very often or always true. The total possible range of scores is 8-40 where higher scores indicate a greater ability to focus.
Time Frame: Baseline, week 1, week 2, week 3, week 4 (of intervention period), and 3 month follow-up
Population: Some participants did not provide data at all time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care
Number analyzed (Participants) | 462 | 463 | 232
score on a scale
  baseline | 24.11 (6.13) | 24.41 (6.32) | 23.95 (6.57)
  Week 1: number analyzed (Participants) | 402 | 407 | 215
  Week 1 | 23.61 (6.88) | 24.26 (6.91) | 24.27 (7.35)
  Week 2: number analyzed (Participants) | 376 | 377 | 204
  Week 2 | 24.55 (7.1) | 25.02 (7.02) | 24.63 (7.29)
  Week 3: number analyzed (Participants) | 371 | 366 | 204
  Week 3 | 25.68 (7.28) | 25.95 (7.4) | 24.74 (7.65)
  Week 4: number analyzed (Participants) | 395 | 389 | 217
  Week 4 | 25.89 (6.74) | 26.03 (6.83) | 24.68 (6.92)
  3-month follow-up: number analyzed (Participants) | 369 | 368 | 203
  3-month follow-up | 26.09 (6.78) | 26.18 (6.32) | 24.75 (6.75)

6. Secondary Outcome: Connection Measured by NIH Toolbox Loneliness Score
Description: The NIH Toolbox Loneliness is a 5-item questionnaire where participants report how often in the past week they have felt loneliness. It is scored on a 5-point Likert scale where 1 = never to 5 = always. The total possible range of scores is 5-25 where higher scores indicate a greater sense of loneliness.
Time Frame: Baseline, week 1, week 2, week 3, week 4 (of intervention period), and 3 month follow-up
Population: Some participants did not provide data at all time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care
Number analyzed (Participants) | 462 | 463 | 232
score on a scale
  baseline | 15.1 (4.85) | 14.74 (4.63) | 15.13 (4.66)
  Week 1: number analyzed (Participants) | 402 | 407 | 215
  Week 1 | 14.33 (5.11) | 13.97 (4.82) | 14.57 (4.81)
  Week 2: number analyzed (Participants) | 376 | 377 | 204
  Week 2 | 13.52 (5.14) | 13.24 (4.64) | 13.86 (4.98)
  Week 3: number analyzed (Participants) | 371 | 366 | 204
  Week 3 | 13.05 (5.28) | 13.00 (4.79) | 14.21 (4.85)
  Week 4: number analyzed (Participants) | 395 | 389 | 217
  Week 4 | 12.54 (5.30) | 12.41 (4.74) | 14.16 (4.73)
  3-month follow-up: number analyzed (Participants) | 369 | 368 | 203
  3-month follow-up | 12.31 (5.11) | 12.82 (4.96) | 14.10 (4.81)

7. Secondary Outcome: Decentering Measured by Decentering Subscale of Experiencing Questionnaire Scale Score
Description: The Decentering subscale of the Experience Questionnaire is an 11-item questionnaire where participants report on their ability to decenter from their experience. It is scored on a 5-point Likert scale where 1 = never to 5 = all the time. The total possible range of scores is 11-55 where higher scores indicate a greater ability to decenter from experience.
Time Frame: Baseline, week 1, week 2, week 3, week 4 (of intervention period), and 3 month follow-up
Population: Some participants did not provide data at all time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care
Number analyzed (Participants) | 462 | 463 | 232
score on a scale
  baseline | 33.12 (6.65) | 33.22 (6.95) | 33.51 (7.40)
  Week 1: number analyzed (Participants) | 401 | 407 | 214
  Week 1 | 34.15 (6.31) | 33.92 (6.42) | 33.99 (6.94)
  Week 2: number analyzed (Participants) | 376 | 377 | 204
  Week 2 | 36.49 (6.14) | 35.74 (6.40) | 34.43 (6.70)
  Week 3: number analyzed (Participants) | 371 | 366 | 203
  Week 3 | 37.46 (6.46) | 36.69 (6.67) | 34.74 (6.65)
  Week 4: number analyzed (Participants) | 395 | 387 | 217
  Week 4 | 39.05 (6.98) | 37.94 (7.17) | 34.67 (6.96)
  3-month follow-up: number analyzed (Participants) | 367 | 367 | 200
  3-month follow-up | 39.26 (7.37) | 38.37 (7.42) | 35.55 (7.04)

8. Secondary Outcome: Meaning in Life Measured by NIH Toolbox Meaning and Purpose Score
Description: The PROMIS / NIH Toolbox Meaning and Purpose is a computer-adaptive measure where participants report how much meaning and purpose they experience in life (e.g., "I understand my life's meaning"). It is scored on a 5-point Likert scale where 1 = strongly disagree to 5 = strongly agree. It provides total scores as T-scores (mean = 50, SD = 10) where higher scores indicate more meaning and purpose in life.
Time Frame: Baseline, week 1, week 2, week 3, week 4 (of intervention period), and 3 month follow-up
Population: Some participants did not provide data at all time points.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care
Number analyzed (Participants) | 462 | 463 | 232
T-score
  baseline | 43.44 (9.89) | 43.09 (9.78) | 43.33 (9.76)
  Week 1: number analyzed (Participants) | 402 | 407 | 215
  Week 1 | 42.89 (9.64) | 42.59 (9.74) | 41.58 (9.67)
  Week 2: number analyzed (Participants) | 376 | 377 | 204
  Week 2 | 44.07 (9.89) | 43.66 (9.96) | 41.71 (11.03)
  Week 3: number analyzed (Participants) | 371 | 366 | 204
  Week 3 | 44.98 (10.25) | 44.27 (10.47) | 41.96 (10.61)
  Week 4: number analyzed (Participants) | 395 | 389 | 217
  Week 4 | 46.86 (11.07) | 45.74 (10.63) | 42.88 (10.47)
  3-month follow-up: number analyzed (Participants) | 368 | 368 | 202
  3-month follow-up | 47.64 (10.93) | 46.19 (10.69) | 44.21 (10.60)

9. Secondary Outcome: Pain Intensity Measured by PROMIS Pain Intensity Score
Description: The single-item PROMIS Pain Intensity scale is a 1-item scale where participants report on their pain intensity in the past 7 days. It is scored on an 11-point Likert-scale where 0 = no pain and 10 = worst pain imaginable. Scores range from 0 to 10, with higher scores indicating higher pain intensity
Time Frame: Baseline, week 4 (of intervention period), and 3 month follow-up
Population: Some participants did not provide data at all time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care
Number analyzed (Participants) | 462 | 463 | 232
score on a scale
  baseline | 3.22 (2.54) | 3.33 (2.53) | 3.42 (2.59)
  Week 4: number analyzed (Participants) | 395 | 389 | 217
  Week 4 | 2.98 (2.6) | 3.12 (2.57) | 3.5 (2.81)
  3-month follow-up: number analyzed (Participants) | 367 | 368 | 201
  3-month follow-up | 3.11 (2.63) | 3.07 (2.59) | 3.39 (2.73)

10. Secondary Outcome: Pain Interference Measured by PROMIS Pain Inference Scale Score
Description: The PROMIS Pain Interference scale is a computer-adaptive measure where participants report how often in the past 7 days they had pain-related interference in their life (e.g., "how much did pain interfere with your enjoyment of life"). It is scored on a 5-point Likert scale where 1 = not at all to 5 = very much. It provides total scores as T-scores (mean = 50, SD = 10) where higher scores indicate more pain interference.
Time Frame: Baseline, week 4 (of intervention period), and 3 month follow-up
Population: Some participants did not provide data at all time points.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care
Number analyzed (Participants) | 462 | 463 | 232
T-score
  baseline | 52.94 (10.27) | 53.6 (10.17) | 53.57 (10.51)
  Week 4: number analyzed (Participants) | 395 | 389 | 217
  Week 4 | 51.65 (10.55) | 51.66 (9.81) | 53.16 (10.91)
  3-month follow-up: number analyzed (Participants) | 368 | 368 | 201
  3-month follow-up | 52.21 (10.65) | 52.13 (10.17) | 52.96 (11.06)

11. Secondary Outcome: Nonjudgment Measured by Five Facet Mindfulness Questionnaire Nonjudgment Subscale Score
Description: The Five Facet Mindfulness Questionnaire Nonjudgment Subscale is a 8-item subscale where participants report on their nonjudgment of experience in daily life. It is scored on a 5-point Likert scale where 1 = never or very rarely true to 5 = very often or always true. The total possible range of scores is 8-40 where higher scores indicate a greater nonjudgment of experience.
Time Frame: Baseline, week 1, week 2, week 3, week 4 (of intervention period), and 3 month follow-up
Population: Some participants did not provide data at all time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care
Number analyzed (Participants) | 462 | 463 | 232
score on a scale
  baseline | 24.62 (7.05) | 24.35 (6.88) | 23.92 (6.89)
  Week 1: number analyzed (Participants) | 402 | 407 | 215
  Week 1 | 26.24 (7.45) | 26.32 (7.47) | 25.84 (7.80)
  Week 2: number analyzed (Participants) | 376 | 377 | 204
  Week 2 | 27.98 (7.46) | 27.46 (7.55) | 26.88 (7.67)
  Week 3: number analyzed (Participants) | 371 | 366 | 204
  Week 3 | 29.53 (7.50) | 28.57 (7.68) | 26.99 (7.97)
  Week 4: number analyzed (Participants) | 395 | 389 | 217
  Week 4 | 28.93 (6.86) | 28.16 (6.90) | 26.35 (7.62)
  3-month follow-up: number analyzed (Participants) | 369 | 368 | 203
  3-month follow-up | 28.89 (6.77) | 27.83 (6.95) | 26.12 (7.42)

12. Secondary Outcome: Climate Change Anxiety Scale
Description: The Climate Change Anxiety Scale is a 13-item scale where participants report their anxiety regarding climate change (e.g., "I have nightmares about climate change"). It is scored on a 5-point Likert scale where 1 = "never" to 5 = "almost always." Total scores range from 13 to 65 where higher scores indicate greater climate change anxiety.
Time Frame: Baseline, week 4, and 3 month follow up
Population: Some participants did not provide data at all time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care
Number analyzed (Participants) | 462 | 463 | 232
score on a scale
  baseline | 21.17 (7.02) | 20.98 (7.54) | 21.22 (7.91)
  Week 4: number analyzed (Participants) | 395 | 387 | 217
  Week 4 | 20.79 (6.95) | 20.67 (7.51) | 21.01 (8.18)
  3-month follow-up: number analyzed (Participants) | 367 | 367 | 200
  3-month follow-up | 20.5 (6.68) | 20.34 (7.74) | 20.18 (8.33)

13. Secondary Outcome: Wellbeing Growth Mindset
Description: The Wellbeing Growth Mindset scale is a 3-item scale where participants report whether they believe wellbeing is malleable (e.g., "Your well-being is something about you that you can't change very much."). It is scored on a 6-point Likert scale where 1 = "strongly disagree" to 6 = "strongly agree." Total scores range from 3 to 18 where higher scores indicate greater wellbeing growth mindset.
Time Frame: Baseline, week 4, and 3 month follow up
Population: Some participants did not provide data at all time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care
Number analyzed (Participants) | 462 | 463 | 232
score on a scale
  baseline | 14.27 (2.83) | 14.07 (2.89) | 13.88 (3.17)
  Week 4: number analyzed (Participants) | 395 | 389 | 218
  Week 4 | 14.61 (2.90) | 14.46 (2.70) | 13.50 (3.23)
  3-month follow-up: number analyzed (Participants) | 371 | 368 | 203
  3-month follow-up | 14.31 (2.93) | 14.04 (3.10) | 13.54 (3.12)

14. Secondary Outcome: Healthy Minds Index (HM Index) - Awareness
Description: The HM Index is a 17-item questionnaire assessing qualities trained in the HMP app (awareness, connection, insight, purpose). It is scored on a 0- to 4-point Likert scale where 0 = a low amount (e.g., never, not at all, none of the time) and 4 = a higher amount (e.g., always, to the highest degree, all of the time) of a particular quality. Total scores for the Awareness subscale is 0 to 16 where higher scores indicate more awareness.
Time Frame: Baseline, week 4, and 3 month follow up
Population: Some participants did not provide data at all time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care
Number analyzed (Participants) | 462 | 463 | 232
score on a scale
  baseline | 9.13 (2.72) | 9.11 (2.8) | 9.01 (2.86)
  Week 4: number analyzed (Participants) | 395 | 389 | 218
  Week 4 | 9.55 (2.75) | 9.33 (2.94) | 8.72 (2.91)
  3-month follow-up: number analyzed (Participants) | 371 | 369 | 203
  3-month follow-up | 9.72 (2.78) | 9.5 (2.88) | 8.89 (2.76)

15. Secondary Outcome: Healthy Minds Index (HM Index) - Connection
Description: The HM Index is a 17-item questionnaire assessing qualities trained in the HMP app (awareness, connection, insight, purpose). It is scored on a 0- to 4-point Likert scale where 0 = a low amount (e.g., never, not at all, none of the time) and 4 = a higher amount (e.g., always, to the highest degree, all of the time) of a particular quality. Total scores for the Connection subscale range from 0 to 24, where higher scores indicate more connection.
Time Frame: Baseline, week 4, and 3 month follow up
Population: Some participants did not provide data at all time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care
Number analyzed (Participants) | 462 | 463 | 232
score on a scale
  baseline | 15.67 (3.79) | 15.65 (3.49) | 15.64 (3.64)
  Week 4: number analyzed (Participants) | 395 | 389 | 218
  Week 4 | 16.03 (4.03) | 16.16 (3.86) | 15.16 (3.72)
  3-month follow-up: number analyzed (Participants) | 371 | 369 | 203
  3-month follow-up | 15.88 (4.02) | 16.03 (3.81) | 15.08 (3.94)

16. Secondary Outcome: Healthy Minds Index (HM Index) - Insight
Description: The HM Index is a 17-item questionnaire assessing qualities trained in the HMP app (awareness, connection, insight, purpose). It is scored on a 0- to 4-point Likert scale where 0 = a low amount (e.g., never, not at all, none of the time) and 4 = a higher amount (e.g., always, to the highest degree, all of the time) of a particular quality. Total scores for the Insight subscale range from 0 to 12, where higher scores indicate more insight.
Time Frame: Baseline, week 4, and 3 month follow up
Population: Some participants did not provide data at all time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care
Number analyzed (Participants) | 462 | 463 | 232
score on a scale
  baseline | 5.79 (2.3) | 5.76 (2.44) | 6.03 (2.24)
  Week 4: number analyzed (Participants) | 395 | 389 | 218
  Week 4 | 6.78 (2.31) | 6.71 (2.29) | 6.07 (2.16)
  3-month follow-up: number analyzed (Participants) | 371 | 369 | 203
  3-month follow-up | 6.86 (2.34) | 6.89 (2.23) | 6.08 (2.26)

17. Secondary Outcome: Healthy Minds Index (HM Index) - Purpose
Description: The HM Index is a 17-item questionnaire assessing qualities trained in the HMP app (awareness, connection, insight, purpose). It is scored on a 0- to 4-point Likert scale where 0 = a low amount (e.g., never, not at all, none of the time) and 4 = a higher amount (e.g., always, to the highest degree, all of the time) of a particular quality. Total scores for the Purpose subscale range from 0 to 16, where higher scores indicate more purpose.
Time Frame: Baseline, week 4, and 3 month follow up
Population: Some participants did not provide data at all time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care
Number analyzed (Participants) | 462 | 463 | 232
score on a scale
  baseline | 9.07 (3.57) | 8.8 (3.71) | 9.22 (3.61)
  Week 4: number analyzed (Participants) | 395 | 389 | 218
  Week 4 | 10.19 (3.47) | 10.05 (3.56) | 8.95 (3.61)
  3-month follow-up: number analyzed (Participants) | 371 | 369 | 203
  3-month follow-up | 10.48 (3.34) | 10.16 (3.56) | 9.43 (3.95)

18. Secondary Outcome: Life Orientation Test - Revised
Description: The Life Orientation Test - Revised is a 6-item scale where participants report their level of optimism (e.g., "In uncertain times, I usually expect the best"). It is scored on a 5-point Likert scale where 0 = "strongly disagree" to 4 = "strongly agree." Total scores range from 0 to 24 where higher scores indicate greater optimism.
Time Frame: Baseline, week 4, and 3 month follow up
Population: Some participants did not provide data at all time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care
Number analyzed (Participants) | 462 | 463 | 232
score on a scale
  baseline | 11.78 (4.97) | 11.71 (4.72) | 11.77 (5.21)
  Week 4: number analyzed (Participants) | 395 | 389 | 217
  Week 4 | 13.42 (5.02) | 13.01 (4.73) | 12.23 (4.98)
  3-month follow-up: number analyzed (Participants) | 368 | 368 | 202
  3-month follow-up | 13.73 (5.13) | 13.17 (4.83) | 12.22 (5.32)

19. Secondary Outcome: Perceived Stress Scale
Description: The Perceived Stress Scale is a 10-item scale where participants report their level of perceived stress (e.g., "In the last month, how often have you felt nervous and 'stressed'?"). It is scored on a 5-point Likert scale where 0 = "never" to 4 = "very often." Total scores range from 0 to 40 where higher scores indicate greater perceived stress.
Time Frame: Baseline, week 4, and 3 month follow up
Population: Some participants did not provide data at all time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care
Number analyzed (Participants) | 462 | 463 | 232
score on a scale
  baseline | 29.7 (6.77) | 29.51 (6.29) | 29.72 (6.64)
  Week 4: number analyzed (Participants) | 395 | 389 | 217
  Week 4 | 26.46 (6.82) | 26.90 (6.54) | 29.17 (6.54)
  3-month follow-up: number analyzed (Participants) | 68 | 368 | 201
  3-month follow-up | 25.70 (7.37) | 26.03 (7.10) | 28.45 (7.11)

20. Secondary Outcome: Perseverative Thinking Questionnaire
Description: The Perseverative Thinking Questionnaire is a 15-item scale where participants report their level of repetitive negative thinking (e.g., "My thoughts repeat themselves"). It is scored on a 5-point Likert scale where 0 = "never" to 4 = "almost always." Total scores range from 0 to 60 where higher scores indicate greater perseverative thinking.
Time Frame: Baseline, week 4, and 3 month follow up
Population: Some participants did not provide data at all time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care
Number analyzed (Participants) | 462 | 463 | 232
score on a scale
  baseline | 32.02 (11.34) | 31.14 (11.56) | 31.56 (11.83)
  4 week: number analyzed (Participants) | 395 | 388 | 217
  4 week | 26.94 (11.90) | 27.08 (11.59) | 30.69 (11.93)
  3-month follow-up: number analyzed (Participants) | 367 | 368 | 200
  3-month follow-up | 25.39 (12.40) | 26.48 (12.03) | 29.28 (12.55)

21. Secondary Outcome: Satisfaction With Life Scale
Description: The Satisfaction with Life Scale is a 5-item scale where participants report their level of satisfaction with life (e.g., "In most ways my life is close to ideal"). It is scored on a 7-point Likert scale where 1 = "strongly disagree" to 7 = "strongly agree." Total scores range from 5 to 35 where higher scores indicate greater satisfaction with life.
Time Frame: Baseline, week 4, and 3 month follow up
Population: Some participants did not provide data at all time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care
Number analyzed (Participants) | 462 | 463 | 232
score on a scale
  baseline | 17.25 (7.30) | 17.27 (7.24) | 17.08 (7.22)
  Week 4: number analyzed (Participants) | 395 | 389 | 217
  Week 4 | 19.62 (7.72) | 19.40 (7.37) | 17.51 (7.47)
  3-month follow-up: number analyzed (Participants) | 368 | 368 | 201
  3-month follow-up | 20.33 (7.81) | 19.94 (7.61) | 18.04 (7.42)

22. Secondary Outcome: Subjective Happiness Scale
Description: The Subjective Happiness Scale is a 4-item scale where participants report their level of subjective happiness (e.g., "In general, I consider myself [not a very happy person, a very happy person]"). It is scored on a 7-point Likert scale where 1 = less happy to 7 = more happy. Total scores range from 4 to 28 where higher scores indicate greater subjective happiness.
Time Frame: Baseline, week 4, and 3 month follow up
Population: Some participants did not provide data at all time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care
Number analyzed (Participants) | 462 | 463 | 232
score on a scale
  baseline | 16.45 (4.96) | 16.53 (5.25) | 16.29 (4.93)
  Week 4: number analyzed (Participants) | 395 | 388 | 217
  Week 4 | 17.91 (5.14) | 17.36 (5.24) | 16.35 (4.94)
  3-month follow-up: number analyzed (Participants) | 367 | 368 | 201
  3-month follow-up | 18.20 (5.31) | 17.77 (5.54) | 16.62 (4.93)

23. Secondary Outcome: Problematic and Risky Internet Use Screening Scale (PRIUSS-3)
Description: The PRIUSS-3 is a 3-item scale where participants report their level of problematic internet use. It is scored on a 4-point Likert scale where 0 = never to 4 = very often. Total scores range from 0 to 12, where higher scores indicate more problematic internet use.
Time Frame: Baseline, week 4, and 3 month follow up
Population: Some participants did not provide data at all time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care
Number analyzed (Participants) | 462 | 463 | 232
score on a scale
  baseline: number analyzed (Participants) | 201 | 202 | 101
  baseline | 4.79 (2.68) | 4.45 (2.74) | 4.42 (2.87)
  Week 4: number analyzed (Participants) | 204 | 191 | 113
  Week 4 | 3.96 (2.83) | 3.97 (2.76) | 4.94 (3.15)
  3-month follow-up: number analyzed (Participants) | 250 | 253 | 136
  3-month follow-up | 3.81 (2.75) | 3.63 (2.61) | 4.50 (2.82)

24. Other Pre Specified Outcome: Inflammatory Biomarkers: C-reactive Protein (CRP)
Description: Dried blood spot samples will be used to measure two inflammatory cytokines (C-reactive protein (CRP) and interleukin-6 (IL-6)). Additionally mRNA assays will be used to detect and quantify inflammatory gene expression detect and monitor cellular immune responses. Analyses will focus on transcripts from ~200 genes known to be involved in the regulation of inflammation, and will consider key transcripts (e.g., IL-1beta, TNF-alpha) as well as summary measures reflecting the activity of transcriptional networks that coordinate inflammation (NF-kB, AP-1).
Time Frame: Baseline and 3 month follow-up
Population: Data not provided or evaluable from all participants at all time points
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care
Number analyzed (Participants) | 462 | 463 | 232
mg/L
  baseline: number analyzed (Participants) | 340 | 341 | 177
  baseline | 2.34 (3.99) | 2.68 (4.16) | 2.67 (2.43)
  3-month follow-up: number analyzed (Participants) | 337 | 338 | 175
  3-month follow-up | 2.56 (4.17) | 2.89 (4.55) | 2.60 (4.05)

25. Other Pre Specified Outcome: Inflammatory Biomarkers: TNF-Alpha, IL-6, Il-10
Description: as for outcome 24
Time Frame: Baseline and 3 month follow-up
Population: Data not provided or evaluable from all participants at all time points
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care
Number analyzed (Participants) | 462 | 463 | 232
pg/mL
  TNF-Alpha at baseline: number analyzed (Participants) | 321 | 328 | 171
  TNF-Alpha at baseline | 2.12 (7.08) | 1.69 (0.85) | 1.75 (0.79)
  TNF-Alpha at 3-month follow-up: number analyzed (Participants) | 321 | 323 | 167
  TNF-Alpha at 3-month follow-up | 1.83 (3.71) | 1.62 (0.83) | 2.02 (3.11)
  IL-6 at baseline: number analyzed (Participants) | 320 | 328 | 171
  IL-6 at baseline | 0.81 (6.94) | 0.33 (0.36) | 0.36 (0.48)
  IL-6 at 3-month follow-up: number analyzed (Participants) | 321 | 323 | 167
  IL-6 at 3-month follow-up | 0.81 (5.18) | 0.37 (0.68) | 0.73 (2.95)
  IL-10 at baseline: number analyzed (Participants) | 321 | 328 | 171
  IL-10 at baseline | 0.12 (0.19) | 0.13 (0.23) | 0.36 (2.76)
  IL-10 at 3-month follow-up: number analyzed (Participants) | 320 | 322 | 167
  IL-10 at 3-month follow-up | 0.13 (0.20) | 0.14 (0.25) | 0.37 (2.81)

26. Other Pre Specified Outcome: Microbiome Alpha Diversity: Species Richness
Description: Genetic analyses of the microbiome of the fecal sample (microorganism DNA, not that of the person) will be performed. Reported here are the observed (total number of distinct taxa) and calculated (Chao1 = N + S2 / (2 D), where N is the number of observed OTUs (Operational Taxonomic Units), S is the number of singleton OTUs, and D is the number of doublet OTUs) number of species represented in the sample. Chao1 is a species richness calculator that accounts for rare species.
Time Frame: Baseline and 3 month follow-up
Population: Some participants did not provide data at all time-points.
Measure: Mean (Standard Deviation); unit: species
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care
Number analyzed (Participants) | 462 | 463 | 232
species
  Observed at baseline: number analyzed (Participants) | 342 | 344 | 176
  Observed at baseline | 308.78 (122.78) | 300.80 (117.87) | 312.68 (114.24)
  Observed at 3-month follow-up: number analyzed (Participants) | 331 | 329 | 174
  Observed at 3-month follow-up | 303.48 (120.49) | 300.88 (116.95) | 311.52 (115.26)
  Calculated at baseline: number analyzed (Participants) | 342 | 344 | 176
  Calculated at baseline | 309.89 (123.30) | 301.88 (118.55) | 313.87 (114.89)
  Calculated at 3-month follow-up: number analyzed (Participants) | 331 | 329 | 174
  Calculated at 3-month follow-up | 304.58 (120.94) | 301.97 (117.57) | 312.64 (115.77)

27. Other Pre Specified Outcome: Microbiome Alpha Diversity: Shannon Diversity Index (H')
Description: Genetic analyses of the microbiome of the fecal sample (microorganism DNA, not that of the person) will be performed. Shannon Diversity Index quantifies both the richness and the evenness of a community. It takes into account the number of taxa (richness) and their relative abundances (evenness). A higher Shannon index value indicates greater diversity, with both a high number of taxa and more even distribution of abundances among them. It is often used to assess the balance between species in a community. Typically ranges from 0-5 with higher numbers indicating increasing species diversity.
Time Frame: Baseline and 3 month follow-up
Population: Some participants did not provide data at all time-points.
Measure: Mean (Standard Deviation); unit: H' index
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care
Number analyzed (Participants) | 462 | 463 | 232
H' index
  baseline: number analyzed (Participants) | 342 | 344 | 176
  baseline | 4.20 (0.56) | 4.19 (0.54) | 4.23 (0.52)
  3-month follow-up: number analyzed (Participants) | 331 | 329 | 174
  3-month follow-up | 4.19 (0.61) | 4.20 (0.51) | 4.24 (0.53)

28. Other Pre Specified Outcome: Microbiome Alpha Diversity: Inverse Simpson (1/D)
Description: Genetic analyses of the microbiome of the fecal sample (microorganism DNA, not that of the person) will be performed. Simpson is the probability that any two microbes are the same species, ranging from 0-1. Inverse Simpson (1 / Simpson) considers both richness and evenness. It places greater weight on the more abundant taxa. A higher inverse Simpson index suggests a more even distribution of taxa, with fewer dominant species. The inverse Simpson index is sensitive to the presence of dominant species and may emphasize diversity loss when one or a few species dominate the community.
Time Frame: Baseline and 3 month follow-up
Population: Some participants did not provide data at all time-points.
Measure: Mean (Standard Deviation); unit: 1/D index
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care
Number analyzed (Participants) | 462 | 463 | 232
1/D index
  baseline: number analyzed (Participants) | 342 | 344 | 176
  baseline | 42.62 (45.06) | 42.54 (45.04) | 43.41 (44.28)
  3-month follow-up: number analyzed (Participants) | 331 | 329 | 174
  3-month follow-up | 43.59 (46.13) | 42.21 (44.66) | 44.43 (46.58)

29. Other Pre Specified Outcome: Microbiome Alpha Diversity: Pielou Evenness Index (J)
Description: Genetic analyses of the microbiome of the fecal sample (microorganism DNA, not that of the person) will be performed. Pielou Evenness Index measures how evenly the individuals are distributed across the taxa in a sample. It is calculated by dividing the Shannon diversity index by the maximum possible value of the Shannon index (which occurs when all taxa are equally abundant). The Pielou index ranges from 0 (no evenness, where one species dominates) to 1 (perfect evenness, where all species are equally abundant).
Time Frame: Baseline and 3 month follow-up
Population: Some participants did not provide data at all time-points.
Measure: Mean (Standard Deviation); unit: J index
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care
Number analyzed (Participants) | 462 | 463 | 232
J index
  baseline: number analyzed (Participants) | 342 | 344 | 176
  baseline | 0.74 (0.07) | 0.74 (0.06) | 0.74 (0.07)
  3-month follow-up: number analyzed (Participants) | 331 | 329 | 174
  3-month follow-up | 0.74 (0.08) | 0.75 (0.06) | 0.75 (0.07)

30. Other Pre Specified Outcome: Microbiome Alpha Diversity: Simpson's Dominance Index (D)
Description: Genetic analyses of the microbiome of the fecal sample (microorganism DNA, not that of the person) will be performed. Simpson's Dominance Index measures the probability that two randomly selected individuals from a community belong to the same species (or taxon). It ranges from 0 to 1, where 0 indicates perfect diversity (no dominance of a single species) and values closer to 1 indicate that one or a few species dominate the community. A lower Simpson's dominance score suggests a more diverse community, while a higher score indicates a community dominated by a few taxa.
Time Frame: Baseline and 3 month follow-up
Population: Some participants did not provide data at all time-points.
Measure: Mean (Standard Deviation); unit: D index
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care
Number analyzed (Participants) | 462 | 463 | 232
D index
  baseline: number analyzed (Participants) | 342 | 344 | 176
  baseline | 0.04 (0.03) | 0.04 (0.02) | 0.03 (0.02)
  3-month follow-up: number analyzed (Participants) | 331 | 329 | 174
  3-month follow-up | 0.04 (0.05) | 0.03 (0.02) | 0.03 (0.02)

31. Other Pre Specified Outcome: Facial Behavior: Cheek Raise Score
Description: Participants provide video recordings of their face while responding to a prompt watching brief videos of positive valence (e.g., baby giggling). Data are reported in Action Unit 6 (AU6) of Facial Action Coding System (FACS). FACS is an anatomically-based system for describing facial movement, breaking facial expressions into individual muscle movements called Action Units (AUs). The scores indicate the intensity of cheek movement (0-100), higher movements indicate more intense movement.
Time Frame: Baseline, week 1, week 2, week 3, week 4 (of intervention period), and 3 month follow-up
Population: Some participants did not provide data at all time-points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care
Number analyzed (Participants) | 462 | 463 | 232
score on a scale
  baseline: number analyzed (Participants) | 387 | 386 | 189
  baseline | 11.92 (15.40) | 12.43 (15.97) | 10.06 (12.86)
  Week 1: number analyzed (Participants) | 313 | 308 | 176
  Week 1 | 9.91 (12.61) | 10.05 (13.39) | 8.55 (11.23)
  Week 2: number analyzed (Participants) | 287 | 273 | 162
  Week 2 | 9.77 (12.25) | 10.64 (12.42) | 7.43 (10.60)
  Week 3: number analyzed (Participants) | 266 | 274 | 156
  Week 3 | 10.15 (12.35) | 10.28 (13.73) | 8.29 (12.43)
  Week 4: number analyzed (Participants) | 294 | 277 | 166
  Week 4 | 10.40 (12.27) | 11.16 (14.54) | 8.58 (10.12)
  3-month follow-up: number analyzed (Participants) | 284 | 252 | 154
  3-month follow-up | 11.57 (13.99) | 10.55 (14.88) | 8.60 (12.84)

32. Other Pre Specified Outcome: Lure Discrimination Task (LDI)
Description: Meditation training has the capacity to normalize the overgeneralized inflexible cognition endemic to depression, which is hypothesized to relate to alterations in the hippocampal-dependent process of pattern separation. The investigators will use a pattern separation task to evaluate hippocampal function. The Lure Discrimination Task (LDI) is the difference between the probability of giving a "Similar" response to the lure items (similar to target items) minus the probability of giving a "Similar" response to the foils (unrelated to target items). Larger differences indicate increased discrimination.
Time Frame: Baseline, week 4 (of intervention period), and 3 month follow-up
Population: Some participants did not provide data at all time-points.
Measure: Mean (Standard Deviation); unit: Lure Discrimination Index
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care
Number analyzed (Participants) | 462 | 463 | 232
Lure Discrimination Index
  baseline: number analyzed (Participants) | 444 | 440 | 220
  baseline | 0.44 (0.20) | 0.42 (0.21) | 0.41 (0.21)
  Week 4: number analyzed (Participants) | 365 | 351 | 194
  Week 4 | 0.47 (0.21) | 0.45 (0.22) | 0.44 (0.21)
  3-month follow-up: number analyzed (Participants) | 338 | 329 | 179
  3-month follow-up | 0.48 (0.20) | 0.46 (0.22) | 0.46 (0.22)

33. Other Pre Specified Outcome: Self-Referential Pronoun Use
Description: Participants provide recordings of their voice while responding to a prompt that asks to share information about their day. These recordings provide the opportunity to explore indicators of self-referent, inflexible, & over-generalized thinking within natural language. Reported here is the "I" self-referential word frequency.
Time Frame: Baseline, week 1, week 2, week 3, week 4 (of intervention period), and 3 month follow-up
Population: Some participants did not provide data at all time-points.
Measure: Mean (Standard Deviation); unit: percent self referential words used
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care
Number analyzed (Participants) | 462 | 463 | 232
percent self referential words used
  Baseline: number analyzed (Participants) | 402 | 403 | 208
  Baseline | 8.75 (3.20) | 8.63 (3.43) | 8.47 (3.46)
  Week 1: number analyzed (Participants) | 342 | 334 | 188
  Week 1 | 8.52 (3.46) | 8.42 (3.48) | 8.75 (2.95)
  Week 2: number analyzed (Participants) | 321 | 304 | 171
  Week 2 | 8.48 (3.35) | 8.08 (3.24) | 8.23 (3.42)
  Week 3: number analyzed (Participants) | 317 | 304 | 171
  Week 3 | 8.47 (3.59) | 8.57 (3.18) | 9.01 (3.31)
  Week 4: number analyzed (Participants) | 336 | 321 | 190
  Week 4 | 8.07 (3.28) | 8.28 (3.46) | 8.81 (3.41)
  3-month follow-up: number analyzed (Participants) | 312 | 306 | 167
  3-month follow-up | 8.44 (3.48) | 8.28 (3.32) | 8.67 (3.35)

34. Other Pre Specified Outcome: Negative Affect Word Use: Negative Sentiment
Description: Participants provide recordings of their voice while responding to a prompt that asks to share information about their day. These recordings provide the opportunity to explore negative affect word use. Data are reported in percentage (0-100) where higher numbers indicate more intense negative sentiment.
Time Frame: Baseline, week 1, week 2, week 3, week 4 (of intervention period), and 3 month follow-up
Population: Some participants did not provide data at all time points.
Measure: Mean (Standard Deviation); unit: percent negative words used
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care
Number analyzed (Participants) | 462 | 463 | 232
percent negative words used
  baseline: number analyzed (Participants) | 402 | 403 | 208
  baseline | 2.94 (1.95) | 3.02 (1.97) | 2.87 (2.03)
  Week 1: number analyzed (Participants) | 342 | 334 | 188
  Week 1 | 2.79 (1.88) | 2.90 (2.05) | 2.86 (1.89)
  Week 2: number analyzed (Participants) | 321 | 304 | 171
  Week 2 | 2.76 (1.84) | 2.82 (1.89) | 2.72 (1.90)
  Week 3: number analyzed (Participants) | 317 | 304 | 174
  Week 3 | 2.53 (1.86) | 2.76 (1.87) | 3.06 (2.03)
  Week 4: number analyzed (Participants) | 336 | 321 | 190
  Week 4 | 2.51 (1.81) | 2.48 (1.79) | 2.77 (2.07)
  3-month follow-up: number analyzed (Participants) | 312 | 306 | 167
  3-month follow-up | 2.72 (1.98) | 2.70 (1.90) | 2.89 (2.10)

35. Other Pre Specified Outcome: Negative Affect Word Use: Positive Sentiment
Description: Participants provide recordings of their voice while responding to a prompt that asks to share information about their day. These recordings provide the opportunity to explore negative affect word use. Data are reported in percentage (0-100) where higher numbers indicate greater positive sentiment.
Time Frame: Baseline, week 1, week 2, week 3, week 4 (of intervention period), and 3 month follow-up
Population: Some participants did not provide data at all time points.
Measure: Mean (Standard Deviation); unit: percent positive sentiment
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care
Number analyzed (Participants) | 462 | 463 | 232
percent positive sentiment
  baseline: number analyzed (Participants) | 402 | 403 | 208
  baseline | 3.12 (2.12) | 3.26 (2.23) | 3.32 (2.19)
  Week 1: number analyzed (Participants) | 342 | 334 | 188
  Week 1 | 3.38 (2.21) | 3.21 (2.18) | 3.33 (2.34)
  Week 2: number analyzed (Participants) | 321 | 304 | 171
  Week 2 | 3.29 (2.02) | 3.48 (2.26) | 3.41 (2.19)
  Week 3: number analyzed (Participants) | 317 | 304 | 174
  Week 3 | 3.52 (2.16) | 3.39 (2.10) | 3.20 (2.22)
  Week 4: number analyzed (Participants) | 336 | 321 | 190
  Week 4 | 3.68 (2.32) | 3.73 (2.26) | 3.47 (2.34)
  3-month follow-up: number analyzed (Participants) | 312 | 306 | 167
  3-month follow-up | 3.45 (2.27) | 3.40 (2.19) | 3.55 (2.59)

36. Other Pre Specified Outcome: Treatment Expectancies
Description: The Treatment Expectancies is a 6-item scale assessing how much participants believed the training program was helpful to them. Items assess how participants think (e.g., "At this point, how logical does the program offered to you seem?") and feel (e.g., "At this point, how much do you really feel that the program helped you to reduce your stress symptoms?"). Items are scored on either a 9-point Likert scale (e.g., 1 = "not at all logical" to 9 = "very logical") or on a percentage ("At the end of the program, how much improvement in your symptoms do you really feel occurred?", 0% to 100%). Higher scores reflect higher treatment expectancies.
Time Frame: 3-month follow-up
Population: The usual care arm was not surveyed for this measure per protocol.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care
Number analyzed (Participants) | 395 | 387 | 0
score on a scale | 35.07 (11.28) | 32.13 (11.98) |

37. Other Pre Specified Outcome: Number of Participants With PHQ-8 Scores That Increased by 5 Points or More Compared to Baseline
Description: The PHQ-8 is an 8-item questionnaire where participants report how often in the past 2 weeks they were bothered by specific problems. Increase in scores indicates increase is depression symptoms.
Time Frame: Week 1, Week 2, Week 3, Week 4, 3-month follow-up
Population: Some participants did not provide data at all time-points.
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care
Number analyzed (Participants) | 462 | 463 | 232
Participants
  Overall (any time point) | 78 | 64 | 44
  Week 1: number analyzed (Participants) | 403 | 407 | 216
  Week 1 | 28 | 27 | 15
  Week 2: number analyzed (Participants) | 376 | 377 | 204
  Week 2 | 27 | 25 | 11
  Week 3: number analyzed (Participants) | 372 | 366 | 204
  Week 3 | 30 | 21 | 14
  Week 4: number analyzed (Participants) | 395 | 389 | 218
  Week 4 | 24 | 21 | 14
  3-month follow-up: number analyzed (Participants) | 374 | 369 | 204
  3-month follow-up | 20 | 20 | 17

38. Other Pre Specified Outcome: Digital Working Alliance Inventory
Description: The Digital Working Alliance Inventory is a 6-item scale where participants report their working alliance with the HMP app (e.g., "The HMP app supports me to overcome challenges"). It is scored on a 7-point Likert scale where 1 = "strongly disagree" to 7 = "strongly agree." Total scores range from 6 to 42 where higher scores indicate greater working alliance.
Time Frame: week 1, week 2, week 3, week 4, and 3-month follow-up
Population: Some participants did not provide data at all time points. The usual care arm was not surveyed for this measure per protocol.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care
Number analyzed (Participants) | 462 | 463 | 0
score on a scale
  Week 1: number analyzed (Participants) | 402 | 407 | 0
  Week 1 | 32.04 (6.35) | 30.65 (6.29) |
  Week 2: number analyzed (Participants) | 376 | 377 | 0
  Week 2 | 32.67 (5.84) | 30.89 (6.89) |
  Week 3: number analyzed (Participants) | 371 | 366 | 0
  Week 3 | 33.37 (6.55) | 31.79 (6.9) |
  Week 4: number analyzed (Participants) | 395 | 387 | 0
  Week 4 | 33.72 (6.75) | 32.25 (7.27) |
  3-month follow-up: number analyzed (Participants) | 367 | 368 | 0
  3-month follow-up | 31.94 (7.51) | 30.89 (7.53) |

39. Other Pre Specified Outcome: Inclusion of Nature in Self
Description: The Inclusion of Nature in Self is a single item measure assessing the degree to which someone views nature as a part of their sense of self. Participants indicate which of a series of overlapping circles most closely resembles nature and their self. More overlapping circles indicate greater inclusion of nature in self.
Time Frame: Baseline, week 4 (of intervention period), and 3 month follow-up
Population: Some participants did not provide data at all-time points.
Measure: Mean (Standard Deviation); unit: overlapping circles
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care
Number analyzed (Participants) | 462 | 463 | 232
overlapping circles
  baseline: number analyzed (Participants) | 461 | 462 | 231
  baseline | 4.06 (1.70) | 4.04 (1.73) | 3.89 (1.72)
  Week 4: number analyzed (Participants) | 394 | 385 | 217
  Week 4 | 4.54 (1.65) | 4.26 (1.74) | 4.02 (1.71)
  3-month follow-up: number analyzed (Participants) | 365 | 366 | 200
  3-month follow-up | 4.41 (1.63) | 4.18 (1.73) | 3.84 (1.71)

40. Other Pre Specified Outcome: Mindfulness Adherence Questionnaire
Description: The Mindfulness Adherence Questionnaire informal practice items are 6-items assessing the application of mindfulness during daily life (e.g., "In your daily life, how much of the time were you practicing being gentle and compassionate toward yourself?"). It is scored on a 7-point Likert scale where 0 = "never" to 6 = "always." Total scores range from 0 to 42 where higher scores indicate greater informal mindfulness practice.
Time Frame: week 1, week 2, week 3, week 4, and 3 month follow up
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care
Number analyzed (Participants) | 462 | 463 | 0
score on a scale
  Week 1: number analyzed (Participants) | 401 | 407 | 0
  Week 1 | 18.48 (6.07) | 18.93 (6.27) |
  Week 2: number analyzed (Participants) | 376 | 377 | 0
  Week 2 | 20.61 (6.15) | 20.35 (6.47) |
  Week 3: number analyzed (Participants) | 370 | 366 | 0
  Week 3 | 21.56 (6.49) | 21.09 (6.48) |
  Week 4: number analyzed (Participants) | 395 | 387 | 0
  Week 4 | 22.22 (6.5) | 21.82 (6.95) |
  3-month follow-up: number analyzed (Participants) | 367 | 367 | 0
  3-month follow-up | 21.87 (7.24) | 21.96 (7.05) |

41. Other Pre Specified Outcome: Change in Pre- and Post-practice Positive Affect
Description: Two items assessing positive affect are scored on a 1- to 7-point Likert scale where 1 = not at all and 7 = very much. Data comes from multiple surveys.
Time Frame: Before and after HMP activities week 1, week 2, week 2, and week 4
Population: The usual care arm was not surveyed for this measure per protocol.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Surveys
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care
Number analyzed (Participants) | 462 | 463 | 0
Number analyzed (Surveys) | 8667 | 9269 | 0
score on a scale
  Change from Before and After Intervention Week 1: number analyzed (Participants) | 386 | 420 | 0
  Change from Before and After Intervention Week 1: number analyzed (Surveys) | 2699 | 3252 | 0
  Change from Before and After Intervention Week 1 | 0.54 (0.99) | 0.35 (0.90) |
  Change from Before and After Intervention Week 2: number analyzed (Participants) | 383 | 397 | 0
  Change from Before and After Intervention Week 2: number analyzed (Surveys) | 2228 | 2280 | 0
  Change from Before and After Intervention Week 2 | 0.44 (0.90) | 0.33 (0.83) |
  Change from Before and After Intervention Week 3: number analyzed (Participants) | 381 | 366 | 0
  Change from Before and After Intervention Week 3: number analyzed (Surveys) | 2127 | 2041 | 0
  Change from Before and After Intervention Week 3 | 0.38 (0.80) | 0.28 (0.76) |
  Change from Before and After Intervention Week 4: number analyzed (Participants) | 339 | 340 | 0
  Change from Before and After Intervention Week 4: number analyzed (Surveys) | 1623 | 1696 | 0
  Change from Before and After Intervention Week 4 | 0.36 (0.85) | 0.24 (0.78) |

42. Other Pre Specified Outcome: Change in Pre- and Post-practice Negative Affect
Description: Two items assessing negative affect are scored on a 1- to 7-point Likert scale where 1 = not at all and 7 = very much. Data comes from multiple surveys.
Time Frame: Before and after HMP activities week 1, week 2, week 2, and week 4
Population: The usual care arm was not surveyed for this measure per protocol.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Surveys
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care
Number analyzed (Participants) | 462 | 463 | 0
Number analyzed (Surveys) | 8667 | 9269 | 0
score on a scale
  Change from Before and After Intervention Week 1: number analyzed (Participants) | 386 | 420 | 0
  Change from Before and After Intervention Week 1: number analyzed (Surveys) | 2699 | 3252 | 0
  Change from Before and After Intervention Week 1 | -0.51 (0.92) | -0.42 (0.95) |
  Change from Before and After Intervention Week 2: number analyzed (Participants) | 383 | 397 | 0
  Change from Before and After Intervention Week 2: number analyzed (Surveys) | 2228 | 2280 | 0
  Change from Before and After Intervention Week 2 | -0.38 (0.88) | -0.29 (0.85) |
  Change from Before and After Intervention Week 3: number analyzed (Participants) | 381 | 366 | 0
  Change from Before and After Intervention Week 3: number analyzed (Surveys) | 2117 | 2041 | 0
  Change from Before and After Intervention Week 3 | -0.30 (0.75) | -0.29 (0.79) |
  Change from Before and After Intervention Week 4: number analyzed (Participants) | 339 | 340 | 0
  Change from Before and After Intervention Week 4: number analyzed (Surveys) | 1623 | 1696 | 0
  Change from Before and After Intervention Week 4 | -0.33 (0.82) | -0.21 (0.80) |

43. Other Pre Specified Outcome: Change in Post-practice Focus
Description: A single item assessing focus during HMP activities is scored on a 1- to 7-point Likert scale where 1 = not at all and 7 = most of the time. Data comes from multiple surveys.
Time Frame: Before and after HMP activities week 1, week 2, week 2, and week 4
Population: Data collected only from HMP arm per protocol.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Surveys
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care
Number analyzed (Participants) | 462 | 0 | 0
Number analyzed (Surveys) | 8663 | 0 | 0
score on a scale
  Week 1: number analyzed (Participants) | 386 | 0 | 0
  Week 1: number analyzed (Surveys) | 2697 | 0 | 0
  Week 1 | 5.93 (1.22) |  |
  Week 2: number analyzed (Participants) | 383 | 0 | 0
  Week 2: number analyzed (Surveys) | 2228 | 0 | 0
  Week 2 | 6.08 (1.14) |  |
  Week 3: number analyzed (Participants) | 381 | 0 | 0
  Week 3: number analyzed (Surveys) | 2116 | 0 | 0
  Week 3 | 6.08 (1.23) |  |
  Week 4: number analyzed (Participants) | 339 | 0 | 0
  Week 4: number analyzed (Surveys) | 1622 | 0 | 0
  Week 4 | 6.21 (1.06) |  |

ADVERSE EVENTS:
Time Frame: data collected up to 4 months on study
Arm/Group | Healthy Minds Program (HMP) App | Psychoeducation App | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/462 | 0/463 | 0/232
Serious Adverse Events (participants affected / at risk) | 0/462 | 0/463 | 0/232
Other Adverse Events (participants affected / at risk) | 78/462 | 64/463 | 44/232
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Healthy Minds Program (HMP) App (N=462) | Psychoeducation App (N=463) | Usual Care (N=232)
Increased Symptoms of Depression (Psychiatric disorders) | 78 | 64 | 44 — Increase in scores PHQ-8 scores indicate increase is depression symptoms. This is the number of participants with increases of 5 points or more.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-01-16): https://cdn.clinicaltrials.gov/large-docs/67/NCT05183867/Prot_SAP_001.pdf
  • Informed Consent Form (2023-12-20): https://cdn.clinicaltrials.gov/large-docs/67/NCT05183867/ICF_000.pdf